CLINICAL TRIAL: NCT01509014
Title: Community Pharmacy Assisting in Total Cardiovascular Health
Acronym: CPATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Saskatchewan (Other)
Collaborators: Ministry of Health, Saskatchewan (Other); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCT00971412; NCT00971412 (obsolete NCT alias)
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Statin Therapy; Adherence
Keywords: Statins; Adherence; Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacy Intervention Arm (Experimental): All patients receiving statins from pharmacies allocated to the pharmacist intervention arm of the study
  Interventions: Behavioral: CPATCH intervention to support statin adherence
- Usual Care (No Intervention): Pharmacies not allocated to the intervention arm will serve as the control. They received no training on the CPATCH intervention and provide usual care to patients at their pharmacy.

INTERVENTIONS:
Behavioral: CPATCH intervention to support statin adherence — Routine identification of new statin users (first year of therapy), consistent assessment of barriers to adherence at every dispensation for these patients, reassurance about efficacy and safety, and proactive response to identified adherence barriers.
  Arms: Pharmacy Intervention Arm

SUMMARY:
Despite proven benefits in reducing morbidity and mortality, many patients become nonadherent to statin therapy within the first year of starting. Due to their accessibility and frequent patient contact, pharmacists are well-positioned to improve medication adherence.

The purpose of this study is to determine whether a simple intervention by community pharmacists can improve statin adherence in new statin users.

ELIGIBILITY:
Inclusion Criteria:

* Pharmacies must fill at least 85 statin prescriptions in a six-week period
* CPATCH intervention was given priority over other study initiatives offered by the pharmacy
* All members of pharmacy staff provided informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Mean statin adherence among all eligible new users of statin medications with at least 6 months of follow-up from index prescription | 6 months
  All statin dispensations are captured by the prescription drug plan database. Mean adherence will be measured using the proportion of days covered (sum of days supply for statin prescriptions during study period divided by the number of days of observation). PDC will be adjusted for any days subject was hospitalized during study period.,

SECONDARY OUTCOMES:
Proportion of new statin users with adherence greater than or equal to 80% | 6 months
Persistence with statin use among patients with a minimum of 12 months of follow-up | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- College of Pharmacy and Nutrition, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Evans CD, Eurich DT, Taylor JG, Remillard AJ, Shevchuk YM, Blackburn DF. A pragmatic cluster randomized trial evaluating the impact of a community pharmacy intervention on statin adherence: rationale and design of the Community Pharmacy Assisting in Total Cardiovascular Health (CPATCH) study. Trials. 2010 Jul 8;11:76. doi: 10.1186/1745-6215-11-76. PMID 20615235